CLINICAL TRIAL: NCT07016191
Title: A Randomized, Double-blinded and Placebo-controlled Study on Super-Oxygenated Water
Brief Title: Effect of Super-Oxygenated Water on Blood Oxygen Saturation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inhale, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Inhale-001
Record Dates: First submitted 2025-05-16; First posted 2025-06-11 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Adult Subject
Keywords: Inhale; Super-oxygenated Water; Superoxygenated Water; Blood Oxygen Saturation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhale Water (Experimental): Participants will ingest 12oz of Inhale Super-Oxygenated water
  Interventions: Other: Ingestion of Water
- Normal Water (Placebo Comparator): Participants will ingest 12oz of Source and Taste-matched normal water
  Interventions: Other: Ingestion of Water

INTERVENTIONS:
Other: Ingestion of Water — Ingestion of Super-Oxygenated or Normal water

SUMMARY:
Therapeutic delivery of additional Oxygen to blood stream via hyperbaric and extracorporeal oxygenation that raises blood Oxygen saturation level, apart from oxygenation in the lungs, is known to induce tissue repair, restore normal body functions and improve survival. Despite the clinical benefits obtained from these interventions, Oxygen supplementation is rather a medically involved process requiring access to specialized equipment including hyperbaric chambers, cardiac catheterization laboratory and extracorporeal oxygenators, and is not generally amenable for everyday use. The current prospective study will evaluate a non-invasive route for Oxygen delivery through ingestion of super-oxygenated water in adult volunteers. The participants will be randomly assigned to one of the two study groups viz. Inhale super-oxygenated water or placebo control normal water at 1:1 ratio. Neither the participants nor the study doctor will know the treatment assignment. Pre- and post-ingestion measurements will be conducted to evaluate effect of super-oxygenated water.

DETAILED DESCRIPTION:
Participants will drink 12 oz of their assigned water (Inhale water or source and taste matched normal water). Baseline blood Oxygen saturation and Heart rate will be measured by a pulse oximeter immediately prior to water ingestion. At one-minute post-ingestion, the blood Oxygen saturation and Heart rate will be measured to compare changes over the baseline. Assessment of Energy level and Brain clarity will be performed as a participant reported outcome measure conducted at pre- and post-ingestion time points through questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Legally adult (18 years of age or older)
* Subject must be willing to review and provide a written informed consent
* Subject must agree to the study procedures including water ingestion, and SPO2 and heart rate measurements

Exclusion Criteria:

* Any active and life-threatening medical condition involving hepatic, renal, cardiac, respiratory, endocrine, or gastrointestinal systems, or any blood disorder in view of the Principal Investigator to confound the study
* Female subjects those are pregnant, nursing or planning to become pregnant
* Subjects receiving any experimental medications or have undergone a major surgical procedure in last 30 days
* Subjects are excluded if they have previously utilized the test article (INHALE superoxygenated water) within the last 24 hours, or have undergone bariatric surgery or have received weight-loss medication
* Subjects with known anemia, hemoglobinopathy or other comorbidity necessitating fluid restriction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-11-26 (Actual); Study Completion 2025-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Nayak, PhD, Study Director
Locations (1):
- The Center For Whole Health, Westlake Village, California, United States

IPD SHARING:
Plan to Share IPD: No
The results will be utilized in business decisions and possible publications. At this point the data may or may not be shared.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 60 subjects were enrolled in the study.
Pre-assignment Details: The 60 enrolled subjects were randomized into two arms consisting of 30 subjects in each arm.
Groups:
- Inhale Super-Oxygenated Water: Participants will ingest one serving of Inhale super-oxygenated water (12 oz).
- Placebo Control: Participants will ingest one serving of a source and taste-matched normal water (12 oz).
Period: Overall Study
Arm/Group | Inhale Super-Oxygenated Water | Placebo Control
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All consented study subjects were included in the analyses.
Groups:
- Inhale Super-Oxygenated Water: Ingestion of Inhale super-oxygenated water
- Placebo Control: Ingestion of source and taste-matched normal water as placebo control
- Total: Total of all reporting groups
Arm/Group | Inhale Super-Oxygenated Water | Placebo Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants] — Participants who are eligible and provide informed consent Population: Intent to treat population
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 25 | 27 | 52
    >=65 years | 5 | 3 | 8
Age, Continuous [Median (Inter-Quartile Range); unit: Year] — Participants who are eligible and provide informed consent Population: Intent to treat population
  Year | 49.5 [38.25 to 58.75] | 43.5 [30.5 to 52.8] | 47 [34.25 to 56.25]
Sex: Female, Male [Count of Participants; unit: Participants] — Participants who are eligible and provide informed consent Population: Intent to treat population
  Participants
    Female | 16 | 14 | 30
    Male | 14 | 16 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Subjects were recruited from the United States America Population: Intent to treat population
  participants
    United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: SpO2 Response Rate
Description: Number of participants who experienced an improvement in post-ingestion SpO2. An increase in post-ingestion SpO2 over the pre-ingestion level in the same subject was considered a response.
Time Frame: From pre-ingestion to post-ingestion of water
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Inhale Super-Oxygenated Water | Placebo Control
Number analyzed (Participants) | 30 | 30
Participants
  Positive Response | 21 (0.5404) | 11 (0.3117)
Statistical Analysis 1: Comparison: Inhale Super-Oxygenated Water vs Placebo Control; Test type: Superiority; p = 0.010, Chi-squared — Proportions were compared using a chi-squared test at the two-sided 5% level

2. Primary Outcome: Heart Rate Response Rate
Description: Number of participants who experienced a reduction in post-ingestion heart rate. A decrease in post-ingestion heart rate over the pre-ingestion level in the same subject was considered a response.
Time Frame: From pre-ingestion to post-ingestion of water
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Inhale Super-Oxygenated Water | Placebo Control
Number analyzed (Participants) | 30 | 30
Participants | 21 (2.603) | 14 (1.347)
Statistical Analysis 1: Comparison: Inhale Super-Oxygenated Water vs Placebo Control; Test type: Superiority; p = 0.067, Chi-squared — Proportions were compared using a chi-squared test at the two-sided 5% level

3. Secondary Outcome: Energy Level Response Rate
Description: Number of participants who reported an improvement in post-ingestion energy level. An increase in post-ingestion energy level over the pre-ingestion level in the same subject was considered a response. Energy level was measured by a participant-reported questionnaire titled "Energy Level and Brain Clarity Assessment" with possible scores ranging from 1 (meaning "very-low") through 10 (meaning "very-high") where higher score indicated a greater energy level.
Time Frame: From pre-ingestion to post-ingestion of water
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Inhale Super-Oxygenated Water | Placebo Control
Number analyzed (Participants) | 30 | 30
Participants | 17 (7.520) | 6 (3.278)
Statistical Analysis 1: Comparison: Inhale Super-Oxygenated Water vs Placebo Control; Test type: Superiority; p = 0.003, Chi-squared — Proportions were compared using a chi-squared test at the two-sided 5% level

4. Secondary Outcome: Brain Clarity Response Rate
Description: Number of participants who reported an improvement in post-ingestion brain clarity. An increase in post-ingestion brain clarity over the pre-ingestion level in the same subject was considered a response. Brain clarity was measured by a participant-reported questionnaire titled "Energy Level and Brain Clarity Assessment" with possible scores ranging from 1 (meaning "very-low") through 10 (meaning "very-high") where higher score indicated a greater brain clarity.
Time Frame: From pre-ingestion to post-ingestion of water
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Inhale Super-Oxygenated Water | Placebo Control
Number analyzed (Participants) | 30 | 30
Participants | 15 (3.827) | 5 (3.519)
Statistical Analysis 1: Comparison: Inhale Super-Oxygenated Water vs Placebo Control; Test type: Superiority; p = 0.006, Chi-squared — Proportions were compared using a chi-squared test at the two-sided 5% level

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from time of consent through post-ingestion time point.
Arm/Group | Inhale Super-Oxygenated Water | Placebo Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2025-01-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT07016191/Prot_002.pdf
  • Statistical Analysis Plan (2025-05-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT07016191/SAP_003.pdf
  • Informed Consent Form (2025-02-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT07016191/ICF_004.pdf